CLINICAL TRIAL: NCT03112694
Title: A Multicenter, Retrospective, Medical Record Review Of The Effectiveness Of Lanreotide Following Treatment With Octreotide In Patients With Neuroendocrine Tumors
Brief Title: Switching From Octreotide to Lanreotide - A Look Back at Patients With Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-US-52030-364
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Data collection — This is a non-interventional study, the decision to prescribe the product would have been taken prior to, and independently from the decision to enrol the patient.

SUMMARY:
The purpose of this study is to understand how people with neuroendocrine tumors respond to treatment with lanreotide after having received treatment with octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 years or older at time of locally advanced or metastatic diagnosis
* Patients with a confirmed diagnosis of locally advanced or metastatic Gastroenteropancreatic neuroendocrine tumour (GEP-NET)
* Patients who switched treatment from long acting octreotide LAR to lanreotide, where both treatments were received for the treatment of locally advanced or metastatic GEP-NET. i. Treatment with long acting octreotide LAR monotherapy for at least 90-days before treatment with lanreotide monotherapy (rescue SSA# use permitted). ii. Treatment with lanreotide monotherapy for at least 90-days after treatment with long acting octreotide monotherapy (rescue SSA# use permitted)

Exclusion Criteria:

* Patients with other malignant disease
* Patients who participated in a concomitant clinical trial related to treatment of GEP-NET
* Patients being treated with a Somatostatin analogue (SSA) in combination with other NET treatments excluding rescue SSA#
* Patients who received other primary treatment (e.g., targeted therapy, chemotherapy) for GEP-NET during the interval between octreotide and lanreotide
* Patients with NET familial genetic syndrome (i.e., MEN1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals and clinics
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 4 months (data collection duration)
  Evaluated as responsive disease (i.e., complete response, partial response), stable disease or progressive disease at the last tumor assessment while on treatment with lanreotide (based on tumor imaging, symptoms, biomarker(s) and/or clinical judgement)

SECONDARY OUTCOMES:
Progression-free survival, after treatment with octreotide | 4 months (data collection duration)
  For evaluating progression-free survival events will include radiographic progression per investigator, biomarker progression per investigator, symptom progression per investigator, and death. Adverse events (AEs) will not be considered as an event.
Duration of response to lanreotide, after treatment with octreotide | 4 months (data collection duration)
  For evaluating duration of response events will include radiographic progression per investigator, biomarker progression per investigator, symptom progression per investigator, AEs, and death. Open ended responses will be reviewed during the analysis and determined to be an eligible "event" or not at that time.
Duration of treatment with octreotide and duration of treatment with lanreotide | 4 months (data collection duration)
  Duration of octreotide treatment assessed as time from start of octreotide treatment to stop of octreotide treatment. Duration of lanreotide treatment assessed as time from lanreotide initiation to end of lanreotide treatment (censored at the date of last administration (+lanreotide frequency) for patients who had ongoing lanreotide treatment).
Severity of Adverse Events | 4 months (data collection duration)
  Summarized separately during treatment with octreotide and during treatment with lanreotide, as available
Reasons for switching from octreotide to lanreotide | 4 months (data collection duration)
  Summarized descriptively
Levels of 5-hydroxyindoleacetic acid (5-HIAA) (urine test or blood test) before treatment with octreotide, during treatment with octreotide and during treatment with lanreotide, as available | 4 months (data collection duration)
  Summarized descriptively
Levels of Chromogranin A (CgA) before treatment with octreotide, during treatment with octreotide and during treatment with lanreotide, as available | 4 months (data collection duration)
  Summarized descriptively
Severity of symptoms (i.e., flushing, diarrhea, dyspnea, abdominal pain, edema, nausea) before treatment with octreotide, during treatment with octreotide, and during treatment with lanreotide, as available | 4 months (data collection duration)
  Proportion of patients reporting each symptom

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- United States (8):
  - Moffitt Cancer Center, Tampa, Florida
  - Cancer Center of Kansas, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - National Transitional Research, East Setauket, New York
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania